CLINICAL TRIAL: NCT01425203
Title: Safety and Efficacy of Boceprevir in Combination With Peginterferon Alfa-2b Plus Ribavirin for Treatment of Chronic Hepatitis C Genotype 1 in Russia: Previously Untreated Patients and Patients Who Failed Prior Treatment With Pegylated-Interferon Plus Ribavirin
Brief Title: The Effect of Boceprevir in Russian Participants Diagnosed With Chronic Hepatitis C Genotype 1 (P08160)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P08160; MK-3034-046 (Other: Merck)
Record Dates: First submitted 2011-08-26; First posted 2011-08-29 (Estimated); Results first posted 2014-08-18 (Estimated); Last update posted 2021-02-08 (Actual); Status verified 2021-01

CONDITIONS: Chronic Hepatitis C Genotype 1
MeSH Terms: interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- RGT BOC + PR (Experimental): Participants received PR for 4 weeks before addition of BOC. Participants then received response guided therapy (RGT) with BOC + PR for up to 32 weeks followed by PBO + PR for up to 20 weeks.
  Interventions: Drug: Boceprevir; Biological: peginterferon alfa-2b; Drug: Ribavirin
- PBO + PR (Control) (Placebo Comparator): Participants received PR for 4 weeks before addition of BOC-matched PBO. Participants then received BOC + PR for up to 44 weeks.
  Interventions: Drug: Placebo; Biological: peginterferon alfa-2b; Drug: Ribavirin
- Crossover Arm (Experimental): Participants randomized to the PBO + PR Control arm who failed the futility rule at treatment week (TW) 12 or 24 were rolled over to the Crossover arm and received BOC + PR.
  Interventions: Drug: Boceprevir; Biological: peginterferon alfa-2b; Drug: Ribavirin

INTERVENTIONS:
Drug: Boceprevir — boceprevir 200-mg capsules, 800 mg 3 times a day (TID), orally (PO)
  Other Names: SCH 503034
  Arms: Crossover Arm; RGT BOC + PR
Drug: Placebo — boceprevir-matched placebo four 200-mg capsules PO TID.
  Arms: PBO + PR (Control)
Biological: peginterferon alfa-2b — peginterferon alfa-2b 1.5 μg/kg/wk subcutaneously (SC)
  Other Names: PegIntron
Drug: Ribavirin — ribavirin (weight-based dosing) 800 to 1400 mg/day PO divided twice daily dose (BID).

SUMMARY:
The purpose of this study is to determine whether Boceprevir (BOC, SCH 503034, MK-3034) in combination with Peginterferon Alfa 2-b (PEG) plus Ribavirin (RBV) [PEG+RBV=PR] is effective in the treatment of chronic hepatitis C (CHC) genotype 1 among the Russian population. The primary hypothesis is that the percentage of participants achieving sustained virologic response in the BOC + PR group is superior to that in the Placebo (PBO) + PR group.

ELIGIBILITY:
Inclusion criteria:

* body weight ≥40 kg and ≤125 kg
* previously documented CHC genotype 1 infection;
* must have a liver biopsy with histology consistent with CHC and no other etiology
* if cirrhosis present, must have an ultrasound within 6 months of the screening visit (or between screening and Day 1) with no findings suspicious for hepatocellular carcinoma (HCC)
* agree to use acceptable methods of contraception with partner
* previously untreated with pegylated-interferon (either alfa-2a or alfa-2b) plus RBV or failing prior treatment with pegylated-interferon (either alfa-2a or alfa-2b) plus RBV

Exclusion criteria:

* co-infected with the human immunodeficiency virus (HIV) or hepatitis B virus (Hepatitis B surface antigen [HBsAg] positive).
* required discontinuation of previous interferon or ribavirin regimen for an adverse event (possibly or probably related)
* treatment with ribavirin within 90 days and any interferon-alpha, based on the amendment, should be within 1 month prior to screening
* treatment with any investigational drug within 30 days of the screening visit in this trial
* evidence of decompensated liver disease including, but not limited to, a history or presence of clinical ascites, bleeding varices, or hepatic encephalopathy
* diabetic and/or hypertensive with clinically significant ocular examination findings
* clinical diagnosis of substance abuse of specified drugs within specified timeframes
* any known pre-existing medical condition that could interfere with the participant's participation in and completion of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2011-11-23 (Actual); Primary Completion 2013-10-21 (Actual); Study Completion 2013-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Isakov V, Nikitin I, Chulanov V, Ogurtsov P, Lukyanova E, Long J, Wahl J, Helmond FA; P08160 Trial Investigators. Boceprevir plus peginterferon/ribavirin for treatment of chronic hepatitis C in Russia. World J Hepatol. 2016 Feb 28;8(6):331-9. doi: 10.4254/wjh.v8.i6.331. PMID 26962399
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=P08160&kw=P08160&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 18 Russian sites recruited participants for this boceprevir (BOC) trial.
Pre-assignment Details: Of 238 randomized participants, 237 received at least 1 dose of peginterferon alpha-2b (PEG) + ribavirin (RBV) [PR] and comprised the Full Analysis Set (FAS). 4 discontinued (DC) treatment during the PR lead-in phase and did not receive BOC or Placebo (PBO). 27 from PBO Arm failed the futility time point and were rolled over into Crossover Phase.
Groups:
- Crossover Arm: Participants randomized to the PBO + PR Control arm who failed the futility rule at treatment week (TW) 12 or 24 were rolled over to the Crossover arm and received BOC + PR for 32 weeks and PR for up to 44 weeks depending on HCV-RNA level assessment at Crossover Weeks 4 and 8.
Period: Treatment Phase
Arm/Group | RGT BOC + PR | PBO + PR (Control) | Crossover Arm
Started | 159 | 79 | 0
Treated (FAS) | 159 | 78 | 0
Completed | 132 | 42 | 0
Not Completed | 27 | 37 | 0
Not completed — DC during PR Lead-in Phase | 3 | 1 | 0
Not completed — Failure at futility timepoint | 8 | 27 | 0
Not completed — Other virologic failure criteria | 5 | 3 | 0
Not completed — Unidentified reasons | 11 | 5 | 0
Not completed — Did not receive treatment | 0 | 1 | 0
Period: Crossover Phase
Arm/Group | RGT BOC + PR | PBO + PR (Control) | Crossover Arm
Started | 0 (Phase only for participants in PBO + PR Control arm who failed futility rule at TW12 or 24) | 0 (Phase only for participants in PBO + PR Control arm who failed futility rule at TW12 or 24) | 27 (Phase only for participants in PBO + PR Control arm who failed futility rule at TW12 or 24)
Completed | 0 | 0 | 21
Not Completed | 0 | 0 | 6
Not completed — Failure at futility timepoint | 0 | 0 | 3
Not completed — Other virologic failure criteria | 0 | 0 | 3
Period: Follow-up Phase
Arm/Group | RGT BOC + PR | PBO + PR (Control) | Crossover Arm
Started | 153 (6 participants who started treatment in RGT BOC + PR arm did not enter follow-up.) | 49 (27 starting treatment in PBO+PR Control arm switched to Crossover arm and 2 did not enter follow-up) | 27 (All participants treated in crossover arm entered follow-up.)
Completed | 153 | 49 | 27
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics were reported only for the Full Analysis Set (FAS), which consisted of all randomized participants who received at least 1 dose of any trial medication (PEG, RBV, or BOC) in the Treatment Phase. The Crossover Arm is not included as these participants originally started the study in the PBO + PR Control Arm at Baseline.
Groups:
- Total: Total of all reporting groups
Arm/Group | RGT BOC + PR | PBO + PR (Control) | Total
Number analyzed (Participants) | 159 | 78 | 237
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (9.8) | 38.1 (10.0) | 38.4 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 33 | 98
  Male | 94 | 45 | 139

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virologic Response At Follow-up Week 24 (SVR24) Among Participants Who Received At Least One Dose of Any Trial Medication (Full Analysis Set Population)
Description: SVR24 was defined as an undetectable plasma Hepatitis C Virus-ribonucleic acid (HCV-RNA) level at Follow-up Week 24 (FW24). If a participant was missing FW24 data and had undetectable HCV-RNA at FW12, the participant was considered a sustained virologic responder.
Time Frame: Follow-up Week 24 (up to 72 weeks)
Population: Full Analysis Set (FAS); all randomized participants who received at least 1 dose of any trial medication (PEG, RBV, or BOC) in the Treatment Phase. Participants in the PBO Control Arm who switched to the Crossover Arm were considered failures for SVR24 in this analysis and are not reported here.
Measure: Number; unit: percentage of participants
Arm/Group | RGT BOC + PR | PBO + PR (Control) | Crossover Arm
Number analyzed (Participants) | 159 | 78 | 0
percentage of participants | 74.8 | 46.2 |
Statistical Analysis 1: Comparison: RGT BOC + PR vs PBO + PR (Control); The primary statistical comparison was conducted on the FAS using the stratified Miettinen and Nurminen method at alpha level of 0.050 adjusted for stratification factors, including IL28B genotype and previous treatment as specified at the time of randomization; Test type: Superiority or Other; p < 0.0001, Miettinen and Nurminen Method — Multiplicity adjustment for controlling type 1 error for the primary comparison was based on the step-down approach; Adjusted Difference in Percentages = 29.2, 95% CI 2-sided [16.4 to 41.5] — The difference, 95% CI and p-value are adjusted by stratification factors of IL-28B genotype and previous treatment, based on the Miettinen & Nurminen method

2. Secondary Outcome: Percentage of Participants Achieving SVR24 Among Participants Who Received At Least One Dose of Experimental Trial Drug (Modified Intent-To-Treat [mITT] Population)
Description: SVR24 was defined as an undetectable plasma HCV-RNA level at FW24. If a participant was missing FW24 data and had undetectable HCV-RNA at FW12, the participant was considered a sustained virologic responder.
Time Frame: Follow-up Week 24 (up to 72 weeks)
Population: mITT population included all randomized participants who received ≥1 dose of experimental trial drug: BOC (for Experimental RGT BOC + PR arm) or Placebo (for PBO + PR Control arm). Participants in the PBO Control Arm who switched to the Crossover Arm were considered failures for SVR24 in this analysis and are not reported here.
Measure: Number; unit: percentage of participants
Arm/Group | RGT BOC + PR | PBO + PR (Control) | Crossover Arm
Number analyzed (Participants) | 156 | 77 | 0
percentage of participants | 76.3 | 46.8 |
Statistical Analysis 1: Comparison: RGT BOC + PR vs PBO + PR (Control); The key secondary statistical comparison was conducted on the mITT using the stratified Miettinen and Nurminen method at alpha level of 0.050 adjusted for stratification factors; Test type: Superiority or Other; p < 0.0001, Miettinen and Nurminen Method — Multiplicity adjustment for controlling type 1 error for key secondary comparison based on a step-down approach. Key-secondary comparison was tested only if statistical significance of primary comparison was met at alpha level of 0.050; Adjusted Difference in Percentages = 30.2, 95% CI 2-sided [17.3 to 42.5] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants Achieving Early Virologic Response (EVR) At Treatment Week (TW) 8
Description: EVR was defined as an undetectable HCV-RNA level at TW 8. This analysis was conducted when all participants had completed 8 weeks of the study or had discontinued prior to TW 8.
Time Frame: Treatment Week 8
Population: Full Analysis Set (FAS); all randomized participants who received at least 1 dose of any trial medication (PEG, RBV, or BOC) in the Treatment Phase. The Crossover arm had zero participants at TW8 since the first opportunity for participants in the PBO + PR Control arm to roll over to the Crossover arm was at TW12.
Measure: Number; unit: percentage of participants
Arm/Group | RGT BOC + PR | PBO + PR (Control) | Crossover Arm
Number analyzed (Participants) | 159 | 78 | 0
percentage of participants | 87.4 | 42.3 |
Statistical Analysis 1: Comparison: RGT BOC + PR vs PBO + PR (Control); The percentage of participants achieving EVR at TW8 was compared using the stratified Miettinen and Nurminen method at alpha level of 0.050 adjusted for stratification factors in the FAS population; Test type: Superiority or Other; p < 0.0001, Miettinen and Nurminen Method; Adjusted Difference in Percentages = 45.6, 95% CI 2-sided [33.2 to 57.0] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: RGT BOC+PR Arm and PBO+PR Arm (not entering Crossover): 1st dose to up to 52 weeks; PBO+PR Arm (entering Crossover): 1st dose to up to 48 weeks; Crossover Arm: 1st crossover dose to up to 48 weeks.
Description: Adverse events (AE) were reported for 237 randomized participants treated during the Treatment Period. AEs were not reported for 1 randomized participant that did not receive treatment in the Treatment Period. AEs for the 27 participants who started at Baseline in the Control Arm and switched to the Crossover Arm were also reported separately.
Arm/Group | RGT BOC + PR | PBO + PR (Control) | Crossover Arm
Serious Adverse Events (participants affected / at risk) | 17/159 | 9/78 | 1/27
Other Adverse Events (participants affected / at risk) | 153/159 | 71/78 | 22/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RGT BOC + PR (N=159) | PBO + PR (Control) (N=78) | Crossover Arm (N=27)
Neutropenia (Blood and lymphatic system disorders) | 11 (14) | 4 (4) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Adverse event (General disorders) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis chronic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RGT BOC + PR (N=159) | PBO + PR (Control) (N=78) | Crossover Arm (N=27)
Anaemia (Blood and lymphatic system disorders) | 75 (105) | 19 (31) | 12 (18)
Leukopenia (Blood and lymphatic system disorders) | 62 (103) | 25 (35) | 6 (8)
Neutropenia (Blood and lymphatic system disorders) | 80 (141) | 29 (45) | 8 (15)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (16) | 5 (7) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 18 (22) | 3 (3) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 11 (13) | 5 (5) | 1 (1)
Nausea (Gastrointestinal disorders) | 39 (59) | 9 (15) | 4 (5)
Vomiting (Gastrointestinal disorders) | 9 (12) | 2 (2) | 1 (1)
Asthenia (General disorders) | 44 (63) | 23 (23) | 4 (18)
Chills (General disorders) | 16 (24) | 2 (2) | 0 (0)
Fatigue (General disorders) | 30 (40) | 11 (18) | 1 (3)
Hyperthermia (General disorders) | 8 (51) | 4 (12) | 0 (0)
Influenza like illness (General disorders) | 39 (356) | 14 (72) | 2 (30)
Injection site erythema (General disorders) | 9 (9) | 2 (2) | 0 (0)
Irritability (General disorders) | 17 (18) | 9 (11) | 1 (2)
Pyrexia (General disorders) | 77 (271) | 36 (124) | 1 (2)
Body temperature increased (Investigations) | 8 (14) | 2 (2) | 1 (3)
Weight decreased (Investigations) | 28 (33) | 9 (9) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 10 (10) | 5 (7) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (16) | 4 (4) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 15 (33) | 7 (8) | 0 (0)
Dizziness (Nervous system disorders) | 9 (9) | 7 (7) | 0 (0)
Dysgeusia (Nervous system disorders) | 59 (69) | 3 (5) | 15 (18)
Headache (Nervous system disorders) | 43 (89) | 25 (51) | 5 (13)
Sleep disorder (Psychiatric disorders) | 2 (2) | 4 (4) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 25 (38) | 12 (14) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (7) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 32 (33) | 16 (16) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 12 (12) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 19 (20) | 5 (6) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 10 (17) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator agrees not to publish or publicly present any interim results of trial without prior written consent of Sponsor. Investigator further agrees to provide to Sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial. Sponsor has right to review and comment with respect to publications, abstracts, slides, data analysis and presentation